CLINICAL TRIAL: NCT03720028
Title: Parent-child Interaction and Communication in Families Who Have a Child With Rett Syndrome or Angelman Syndrome
Brief Title: Angelman & Rett Syndrome: Interaction and Communication
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: Snummer
Record Dates: First submitted 2018-10-23; First posted 2018-10-25 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2018-10

CONDITIONS: Behavior, Child; Parent-Child Relations; Communication
MeSH Terms: conditions — Child Behavior; Communication | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Child w Angelman/Rett syndrome: Children with Angelman or Rett syndrome, up to 14 years of age
  Interventions: Behavioral: Observation
- Parent: Parents of Children with Angelman or Rett syndrome
  Interventions: Behavioral: Parental experiences

INTERVENTIONS:
Behavioral: Observation — Describe communication and sensory profile using standardized tests and observations.
  Groups: Child w Angelman/Rett syndrome
Behavioral: Parental experiences — Survey parents' experiences with parent-child interaction and augmentative and alternative communication.
  Groups: Parent

SUMMARY:
We aim to describe the communicative and sensory profile of children with Angelman syndrome or Rett syndrome and their use of augmentative and alternative communication. In addition, parents are surveyed regarding parent-child interaction and access to communication support.

ELIGIBILITY:
Inclusion Criteria:

* Angelman or Rett syndrome

Exclusion Criteria:

* none

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with complex communication needs.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Communication profile | 1 day One-time measurement
  Scores on language tests
Parent interaction | 1 day One-time measurement
  Scores on social tests

CONTACTS AND LOCATIONS:
Locations (1):
- Katholieke Universiteit Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No